CLINICAL TRIAL: NCT00749385
Title: A Randomized, Open-Label, 4-Way Crossover Study to Evaluate Naproxen and Esomeprazole Plasma Levels in Healthy Subjects Following Oral Administration of PN 400, Enteric-Coated Naproxen 500mg Plus Enteric-Coated Esomeprazole 20mg, Enteric-Coated Naproxen 500mg Alone, and Enteric-Coated Esomeprazole 20mg Alone.
Brief Title: A Pharmacokinetic (PK) Study Evaluating Naproxen and Esomeprazole Plasma Levels
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: POZEN (Industry)
Responsible Party: David Taylor, POZEN
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PN400-114
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Last update posted 2008-12-23 (Estimated); Status verified 2008-12

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis | interventions — Naproxen; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): PN 400
  Interventions: Drug: PN 400
- 2 (Active Comparator): Enteric-coated naproxen tablet (500mg) plus enteric-coated esomeprazole capsule(20mg)
  Interventions: Drug: EC naproxen plus EC esomeprazole
- 3 (Active Comparator): Enteric-coated naproxen tablet (500mg)
  Interventions: Drug: EC naproxen
- 4 (Active Comparator): EC esomeprazole capsule (20mg)
  Interventions: Drug: EC esomeprazole

INTERVENTIONS:
Drug: PN 400 — A single tablet containing delayed-release naproxen (500mg) plus immediate-release esomeprazole (20mg)
  Arms: 1
Drug: EC naproxen plus EC esomeprazole — Enteric-coated naproxen tablet (500mg) plus enteric-coated esomeprazole capsule (20mg)
  Other Names: EC Naprosyn and Nexium
  Arms: 2
Drug: EC naproxen — Enteric-coated naproxen tablet (500mg)
  Other Names: EC Naprosyn
  Arms: 3
Drug: EC esomeprazole — Enteric-coated esomeprazole capsule (20mg)
  Other Names: Nexium
  Arms: 4

SUMMARY:
A pharmacokinetic study evaluating naproxen and esomeprazole blood levels in 4 treatments, each containing one or both components.

DETAILED DESCRIPTION:
This study is being conducted to assess the relative bioavailability of naproxen and esomeprazole from a single dose of PN 400 (delayed-release naproxen 500mg / immediate-release esomeprazole 20mg), enteric-coated naproxen 500mg co-administered with enteric-coated esomeprazole 20mg, enteric-coated naproxen 500mg administered alone, and enteric-coated esomeprazole 20mg administered alone.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and non-pregnant, non-lactating females who are either of non-childbearing potential or using an acceptable method of birth control.

Exclusion Criteria:

* Standard exclusion criteria for a study of this nature - no significant medical conditions that might affect the interpretation of the PK data or compromise the safety of the subject.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To assess the single-dose pharmacokinetics and relative bioavailability of esomeprazole in PN 400 (naproxen 500mg / esomeprazole 20mg), the enteric-coated (EC) naproxen 500mg plus EC esomeprazole 20mg and the EC esomeprazole 20mg alone treatments | 12-72 hour PK assessments

SECONDARY OUTCOMES:
To assess the single-dose pharmacokinetics and relative bioavailability of naproxen in PN 400 (naproxen 500mg / esomeprazole 20mg, the EC naproxen 500mg plus EC esomeprazole 20mg, and the EC naproxen 500mg alone treatments. | 72-hour PK assessments
To evaluate the safety of each of the single-dose treatments | Entire study duration (48 days)

CONTACTS AND LOCATIONS:
Locations (1):
- PPD, Austin, Texas, United States